CLINICAL TRIAL: NCT01153711
Title: Relative Bioavailability of 10 mcg Olodaterol (Solution for Inhalation Administered With the Respimat) at Steady State Alone or in Combination With Multiple Doses of 400 mg q.d. Ketoconazole (Tablet) in Healthy Male and Female Volunteers (an Open Label, Fixed Sequence, Phase I Study)
Brief Title: Relative Bioavailability of of Olodaterol and Ketoconazole
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Boehringer Ingelheim, Study Chair, Boehringer Ingelheim
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1222.47; 2010-018527-25 (EudraCT Number: EudraCT)
Record Dates: First submitted 2010-06-29; First posted 2010-06-30 (Estimated); Results first posted 2014-04-30 (Estimated); Last update posted 2014-04-30 (Estimated); Status verified 2014-03

CONDITIONS: Healthy; Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — olodaterol; Ketoconazole

ARMS (2):
- BI 1744 10 mcg (Experimental): solution for oral inhalation
  Interventions: Drug: BI 1744; Drug: Ketoconazole
- Ketoconazole 400 mg (Experimental): tablet
  Interventions: Drug: BI 1744; Drug: Ketoconazole

INTERVENTIONS:
Drug: BI 1744 — 10 mcg solution for oral inhalation
  Arms: Ketoconazole 400 mg
Drug: BI 1744 — 10 mcg solution for oral inhalation
  Arms: BI 1744 10 mcg
Drug: Ketoconazole — 400 mg tablet
  Arms: Ketoconazole 400 mg
Drug: Ketoconazole — 400 mg tablet
  Arms: BI 1744 10 mcg

SUMMARY:
This clinical trial is intended to investigate a possible effect of the p-gp inhibitor ketoconazole on the bioavailability of olodaterol

ELIGIBILITY:
Inclusion criteria Healthy male and female volunteers

Exclusion criteria

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2010-05; Primary Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1222.47.1 Boehringer Ingelheim Investigational Site, Ingelheim, Germany

RESULTS

PARTICIPANT FLOW:
Groups:
- Overall Study: Total number of patients treated in the study. This was an open-label, fixed sequence, phase I trial in healthy volunteers. 32 subjects received in period 1 Olodaterol 10 microgram delivered by Respimat inhaler once daily for 8 days and in period 2 Olodaterol 10 microgram delivered by Respimat inhaler once daily plus 1 tablet Ketoconazole 400mg once daily, both for 14 days.
Period: Overall Study
Arm/Group | Overall Study
Started | 32
Completed | 32
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Overall Study
Number analyzed (Participants) | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.5 (7.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 20

OUTCOME MEASURES:

1. Primary Outcome: Area Under Curve From 0 to 1 Hour at Steady State (AUC0-1,ss)
Description: AUC0-1,ss represents the area under the concentration curve of olodaterol in plasma from 0 to time t=1 hour at steady state, where t is defined as the latest time-point where at least 2/3 of the subjects in both treatment periods reveal quantifiable plasma concentrations of olodaterol. The geometric mean is actually the adjusted geometric mean. The geometric coefficient of variation (gCV) is the intra-individual gCV.
Time Frame: Day 8 of period 1 and day 14 of period 2
Population: Pharmacokinetic (PK) analysis set includes all evaluable subjects in the treated set providing at least 1 observation for at least 1 PK endpoint without important protocol violations.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Picogram*hours/milliliter
Groups:
- Olodaterol: Oral inhalation of Olodaterol 10 microgram solution with Respimat A5 device once daily for 8 days.
- Olodaterol Plus Ketoconazole: Oral inhalation of Olodaterol 10 microgram solution with Respimat A5 device once daily for 14 days plus Ketoconazole 400mg tablet administered orally once daily for 14 days.
Arm/Group | Olodaterol | Olodaterol Plus Ketoconazole
Number analyzed (Participants) | 24 | 31
Picogram*hours/milliliter | 2.512 (16.4) | 4.231 (16.4)
Statistical Analysis 1: Comparison: Olodaterol vs Olodaterol Plus Ketoconazole; Ratio Olodaterol plus Ketoconazole and Olodaterol; Test type: Non-Inferiority or Equivalence — Relative bioavailability; p = 1.0000, ANOVA — P-value for ratio outside interval 0.8-1.25; Adjusted geometric mean ratio; Adjusted geometric mean ratio = 168.4, 90% CI 2-sided [155.5 to 182.4], Standard Deviation 16.4 — The standard deviation is actually the geometric coefficient of variation

2. Primary Outcome: Maximum Concentration at Steady State (Cmax,ss)
Description: Cmax,ss represents the maximum concentration of olodaterol and olodaterol glucuronide in plasma at steady state. The geometric mean is actually the adjusted geometric mean. The geometric coefficient of variation (gCV) is the intra-individual gCV.
Time Frame: Day 8 of period 1 and day 14 of period 2
Population: PK analysis set with evaluable data for this endpoint.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Picogram/milliliter
Arm/Group | Olodaterol | Olodaterol Plus Ketoconazole
Number analyzed (Participants) | 32 | 32
Picogram/milliliter
  Olodaterol (N=26;31) | 3.113 (16.8) | 5.169 (16.8)
  Olodaterol glucuronide (N=32;32) | 5.125 (14.7) | 5.465 (14.7)
Statistical Analysis 1: Comparison: Olodaterol vs Olodaterol Plus Ketoconazole; Ratio Olodaterol plus Ketoconazole and Olodaterol for the category Olodaterol; Test type: Non-Inferiority or Equivalence — Relative bioavailability; p = 1.0000, ANOVA — P-value for ratio outside 0.8-1.25; Adjusted geometric mean ratio; Adjusted geometric mean ratio = 166.1, 90% CI 2-sided [153.6 to 179.6], Standard Deviation 16.8 — The standard deviation is actually the geometric coefficient of variation
Statistical Analysis 2: Comparison: Olodaterol vs Olodaterol Plus Ketoconazole; Ratio Olodaterol plus Ketoconazole and Olodaterol for the category Olodaterol glucuronide; Test type: Non-Inferiority or Equivalence — Relative bioavailability; p = 0.0001, ANOVA — P-value for ratio outside 0.8-1.25; Adjusted geometric mean ratio; Adjusted geometric mean ratio = 106.63, 90% CI 2-sided [100.211 to 113.463], Standard Deviation 14.7 — The standard deviation is actually the geometric coefficient of variation

3. Secondary Outcome: Time From Dosing to the Maximum Concentration at Steady State (Tmax,ss)
Description: tmax,ss represents the time from dosing to maximum concentration of olodaterol and olodaterol glucuronide in plasma at steady state.
Time Frame: Day 8 of period 1 and day 14 of period 2
Population: PK analysis set with evaluable data for this endpoint.
Measure: Median (Full Range); unit: Hours
Arm/Group | Olodaterol | Olodaterol Plus Ketoconazole
Number analyzed (Participants) | 32 | 32
Hours
  Olodaterol (N=26;31) | 0.250 [0.0830 to 0.750] | 0.333 [0.167 to 0.750]
  Olodaterol glucuronide (N=32;32) | 4.00 [1.00 to 12.0] | 3.01 [1.00 to 23.0]

4. Secondary Outcome: Fraction of Urine Excretion From 0 to 24 Hours at Steady State (fe0-24,ss)
Description: fe0-24,ss represents the fraction of olodaterol eliminated in urine from time point 0 to 24 hours after administration at steady state.
Time Frame: Day 8 of period 1 and day 14 of period 2
Population: PK analysis set with evaluable data for this endpoint.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percentage
Arm/Group | Olodaterol | Olodaterol Plus Ketoconazole
Number analyzed (Participants) | 32 | 32
Percentage | 4.29 (35.2) | 6.19 (35.9)

5. Secondary Outcome: Amount of the Analyte Excreted in Urine From 0 to 24 Hours at Steady State (Ae0-24,ss)
Description: Ae0-24,ss represents the amount of olodaterol and olodaterol glucuronide that is eliminated in urine from the time 0 to 24h after administration at steady state. The geometric mean is actually the adjusted geometric mean. The geometric coefficient of variation (gCV) is the intra-individual gCV.
Time Frame: Day 8 of period 1 and day 14 of period 2
Population: PK analysis set with evaluable data for this endpoint.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng
Arm/Group | Olodaterol | Olodaterol Plus Ketoconazole
Number analyzed (Participants) | 32 | 32
ng
  Olodaterol | 428.972 (17.8) | 618.716 (17.8)
  Olodaterol glucuronide | 445.266 (18.9) | 591.620 (18.9)
Statistical Analysis 1: Comparison: Olodaterol vs Olodaterol Plus Ketoconazole; Ratio Olodaterol plus Ketoconazole and Olodaterol for the category Olodaterol; Test type: Non-Inferiority or Equivalence — Relative bioavailability; p = 0.9986, ANOVA — P-value for ratio outside 0.8-1.25; Adjusted geometric mean ratio; Adjusted geometric mean ratio = 144.23, 90% CI 2-sided [133.853 to 155.417], Standard Deviation 17.8 — The standard deviation is actually the geometric coefficient of variation
Statistical Analysis 2: Comparison: Olodaterol vs Olodaterol Plus Ketoconazole; Ratio Olodaterol plus Ketoconazole and Olodaterol for the category Olodaterol glucuronide; Test type: Non-Inferiority or Equivalence — Relative bioavailability; p = 0.8991, ANOVA — P-value for ratio outside 0.8-1.25; Adjusted geometric mean ratio; Adjusted geometric mean ratio = 132.87, 90% CI 2-sided [122.732 to 143.843], Standard Deviation 18.9 — The standard deviation is actually the geometric coefficient of variation

6. Secondary Outcome: Area Under Curve From 0 to 8 Hours at Steady State (AUC0-8,ss)
Description: AUC0-8,ss represents the area under the concentration curve of olodaterol glucuronide in plasma from 0 to time t=8 at steady state, where t is defined as the latest time-point where at least 2/3 of the subjects in both treatment periods reveal quantifiable plasma concentrations of the analyte. The geometric mean is actually the adjusted geometric mean. The geometric coefficient of variation (gCV) is the intra-individual gCV.
Time Frame: Day 8 of period 1 and day 14 of period 2
Population: PK analysis set with evaluable data for this endpoint.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Picogram*hours/milliliter
Arm/Group | Olodaterol | Olodaterol Plus Ketoconazole
Number analyzed (Participants) | 25 | 30
Picogram*hours/milliliter | 27.868 (17.9) | 28.076 (17.9)
Statistical Analysis 1: Comparison: Olodaterol vs Olodaterol Plus Ketoconazole; Ratio Olodaterol plus Ketoconazole and Olodaterol; Test type: Non-Inferiority or Equivalence — Relative bioavailability; p = 0.0001, ANOVA — P-value for ratio outside interval 0.8-1.25; Adjusted geometric mean ratio; Adjusted geometric mean ratio = 100.75, 90% CI 2-sided [92.534 to 109.692], Standard Deviation 17.9 — The standard deviation is actually the geometric coefficient of variation

7. Secondary Outcome: Clinical Relevant Abnormalities for Vital Signs, Blood Chemistry, Haematology, Urinalysis and ECG
Description: Clinical relevant abnormalities for Vital Signs, Blood Chemistry, Haematology, Urinalysis and ECG. New abnormal findings or worsening of baseline conditions were reported as treatment-induced Adverse Events.
Time Frame: First administration of trial medication until 6 days after last administration of trial medication
Population: Treated set (TS) - Treated set includes all patients who were dispensed trial medication and were documented to have taken at least 1 dose of investigational treatment.
Measure: Number; unit: participants
Arm/Group | Olodaterol | Olodaterol Plus Ketoconazole
Number analyzed (Participants) | 32 | 32
participants | 0 | 0

8. Secondary Outcome: Assessment of Tolerability by the Investigator
Description: The investigator assessed tolerability based on adverse events and the laboratory evaluation at the end-of-trial examination. The investigator classified the overall tolerability according to the categories 'good', 'satisfactory', 'not satisfactory', and 'bad'.
Time Frame: End of period 1 and end of period 2
Population: TS
Measure: Number; unit: participants
Arm/Group | Olodaterol | Olodaterol Plus Ketoconazole
Number analyzed (Participants) | 32 | 32
participants
  Good | 32 | 32
  Satisfactory | 0 | 0
  Not satisfactory | 0 | 0
  Bad | 0 | 0
  Not assessable | 0 | 0

ADVERSE EVENTS:
Time Frame: First administration of trial medication until 6 days after last administration of trial medication
Arm/Group | Olodaterol | Olodaterol Plus Ketoconazole
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/32
Other Adverse Events (participants affected / at risk) | 5/32 | 9/32
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Olodaterol (N=32) | Olodaterol Plus Ketoconazole (N=32)
Diarrhoea (Gastrointestinal disorders) | 0 | 2
Dry mouth (Gastrointestinal disorders) | 1 | 2
Nausea (Gastrointestinal disorders) | 0 | 5
Allergy to arthropod bite (Immune system disorders) | 2 | 0
Headache (Nervous system disorders) | 2 | 1
Tremor (Nervous system disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.